CLINICAL TRIAL: NCT05055349
Title: "Comparison Between Intrastromal Corneal Ring Segments and Toric Phakic Posterior Intra-ocular Lenses Implantation in Keratoconus"
Brief Title: Intrastromal Corneal Ring Segments and Toric Phakic Posterior Intra-ocular Lenses Implantation in Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Khalafallah, Principal Investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 324 : 11/2019
Record Dates: First submitted 2021-03-25; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corneal collagen cross linking and intrastromal corneal keraring segments. (Active Comparator): 20 eyes will undergo corneal collagen cross linking (epithelium off) 1 month after Femtosecond laser assisted intrastromal corneal keraring segments
  Interventions: Other: corneal ring segments
- toric phakic posterior IOL implantation and corneal collagen cross linking (Active Comparator): 20 eyes will undergo toric phakic posterior IOL implantation 1 year after corneal collagen cross linking (epithelium off).
  Interventions: Other: corneal ring segments

INTERVENTIONS:
Other: corneal ring segments — ring hard segments inserted within corneal stroma using femtolaser
  Other Names: toric phakic posterior IOL implantation/ corneal collagen cross linking

SUMMARY:
To compare visual and refractive measurements of intrastromal corneal ring segments versus toric phakic posterior intra-ocular lenses implantation in keratoconus

DETAILED DESCRIPTION:
* The study is a prospective comparative interventional case series. It will be conducted in Minia university hospital and Roaa Laser Vision Correction Center.
* Fourty eyes will be evenly allocated into two groups:

Group (A): 20 eyes will undergo corneal collagen cross linking (epithelium off) 1 month after Femtosecond laser assisted intrastromal corneal keraring segments.

Group (B): 20 eyes will undergo toric phakic posterior IOL implantation 1 year after corneal collagen cross linking (epithelium off).

• An informed written consent to be involved in the study will be obtained from each patient.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus grade I to III according to the Amsler-Krumeich classification

Exclusion Criteria:

* Acute hydrops or grade IV keratoconus
* Any ocular diseases or surgeries
* Corneal thickness less than 400 µm at the thinnest corneal point, and at least 450 µm at the incision site for ICRS group
* Corneal pacities

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-22 (Estimated)

PRIMARY OUTCOMES:
pentacam readings | 1 month
  a device that read topometric corneal data and other data

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Khalafallah, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No